CLINICAL TRIAL: NCT03478735
Title: Ultrasound-guided Greater Occipital Nerve Block at the C2 Level Compared to Landmark-based Greater Occipital Nerve Block: A Randomized Controlled Trial
Brief Title: Ultrasound Greater Occipital Nerve Block at C2 Level Compared to Landmark-based Greater Occipital Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew Pingree, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-002724
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Occipital Neuralgia; Cervicogenic Headache; Migraine Without Aura
MeSH Terms: conditions — Post-Traumatic Headache; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided GON Block at C2 (Experimental): Ultrasound Guided Greater Occipital Nerve Block at C2
  Interventions: Procedure: Ultrasound Guided Greater Occipital Nerve Block at C2
- Landmark based GON Block (Active Comparator): Landmark-Based Greater Occipital Nerve Block
  Interventions: Procedure: Landmark-Based Greater Occipital Nerve Block

INTERVENTIONS:
Procedure: Ultrasound Guided Greater Occipital Nerve Block at C2 — Ultrasound guided injection
  Arms: Ultrasound Guided GON Block at C2
Procedure: Landmark-Based Greater Occipital Nerve Block — Traditional landmark-guided technique at the superior nuchal line. This approach relies solely on superficial bone-based anatomic landmarks to infiltrate local anesthetic and corticosteroid around the nerve at the level of the superior nuchal line.
  Arms: Landmark based GON Block

SUMMARY:
This study will compare the analgesic benefit of a traditional landmark-guided GON block with the ultrasound-guided approach over a four week period in patients with occipital neuralgia or cervicogenic headache.

DETAILED DESCRIPTION:
Hypothesis: A novel ultrasound-guided greater occipital nerve (GON) block at the level of C2 will result in significantly lower pain scores after 4 weeks when compared with a traditional landmark-guided approach at the superior nuchal line.

The greater occipital nerve (GON) has been implicated in several conditions that prompt referral to pain medicine specialists, including occipital neuralgia and cervicogenic headache. According to the International Headache Society, a local anesthetic block of the GON can aid in the diagnosis and treatment of occipital neuralgia. Many practitioners perform GON injections using a conventional approach, relying solely on superficial bone-based anatomic landmarks to infiltrate local anesthetic and corticosteroid around the nerve at the level of the superior nuchal line. The ambiguity of these injections poses a risk of anesthetizing adjacent structures or injecting into vessels, such as the occipital artery.

In an attempt to mitigate these risks and improve the efficacy of GON injections, ultrasound has been increasingly utilized. Multiple studies have demonstrated successful ultrasound-guided GON blockade at the superior nuchal line and improvement in pain scores compared to non-guided injections. The investigators' preliminary data confirms the feasibility, efficacy, and safety of an ultrasound-guided GON block technique at the level of C2, but it is not yet known whether this technique provides greater pain relief and functional outcomes compared to traditional injections.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral or bilateral headache symptoms attributed to occipital neuralgia or cervicogenic headache as defined by the International Headache Society's International Classification of Headache Disorders (3rd edition beta version)
2. Age 18 years and older (no upper age limit defined)
3. Imaging of cervical spine within last year (either x-ray, MRI or CT)

Exclusion Criteria:

1. History of cervical spine surgery, trauma, or surgical procedure involving head or neck during the last year
2. Use of new preventative medications 1 month prior or during study enrollment
3. Evidence of impaired sensation in the GON dermatome region (posterior scalp to the vertex of the cranium) from neurological, dermatological, or other disease process
4. Evidence of cranial defect or other anatomical abnormality near the target injection site
5. History of bleeding diathesis, coagulopathy, or current use of anticoagulant medications
6. Pregnancy
7. History of adverse reaction or allergy to local anesthetic agents or corticosteroids
8. Occipital nerve block within the past three months.
9. Unavailability for appropriate follow-up throughout the whole duration of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale (NRS) Pain Score | baseline, 4 weeks
  Pain intensity will be assessed using a NRS marked from 0-10 with fixed intervals, with 0=no pain, and 10=worst pain.

SECONDARY OUTCOMES:
Change in number of patients with medication overuse | baseline, 4 weeks
  The subjects will be provided a headache journal to record the number of days they have been using each of their analgesic medications. Medication overuse will be defined as the use of acetaminophen or non-steroidal anti-inflammatory drugs > 14 days a month, triptan, ergotamine, or combination-analgesic medications (e.g.,caffeine containing) medications >9 days a month, and opioid or butalbital containing medications >5 days a month.
Change in number of headache days per month | baseline, 4 weeks
  The number of headache days per month will be obtained at baseline prior to injection in the pain clinic and at 4 weeks post-injection via telephone.
Change in Headache Impact Test (HIT-6) Score | baseline, 4 weeks
  The HIT-6 show the effect that headaches have on normal daily life and the subject's ability to function. It consists of 6 questions; possible responses being never (6 points each), rarely (8 points each), sometimes (10 points each), very often (11 points each), and always (13 points each). The total score ranges from 36 (little to no impact) to 78 (very severe impact).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Pingree, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials